CLINICAL TRIAL: NCT02257242
Title: BrUOG 326: A Phase I Dose-Escalation Study of Vincristine Sulfate Liposome Injection (Marqibo®) in Combination With Bendamustine and Rituximab (BRiM) in Indolent Non-Hodgkin Lymphoma
Brief Title: Vincristine Sulfate Liposome Injection (Marqibo®), Bendamustine and Rituximab-Phase I Trial in Indolent B-cell Lymphoma
Acronym: BRiM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Spectrum Pharmaceuticals, Inc (Industry); Rhode Island Hospital (Other); The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 326
Record Dates: First submitted 2014-09-30; First posted 2014-10-06 (Estimated); Results first posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-05

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, Small-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone
Keywords: Bendamustine; Rituximab; Vincristine sulfate; Vincristine sulfate liposome injection; Phase I; Escalation With Overdose Control
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab; Bendamustine Hydrochloride; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Vincristine sulfate liposome injection 1.8 mg/m^2 (Experimental): Treatment with the combination of rituximab, bendamustine and vincristine sulfate liposome injection will be repeated every 4 weeks for a maximum of 6 cycles. Dose-limiting toxicities will be evaluated during the first cycle of therapy.
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Vincristine sulfate liposome injection
- Vincristine sulfate liposome injection 1.95 mg/m^2 (Experimental): Treatment with the combination of rituximab, bendamustine and vincristine sulfate liposome injection will be repeated every 4 weeks for a maximum of 6 cycles. Dose-limiting toxicities will be evaluated during the first cycle of therapy.
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Vincristine sulfate liposome injection
- Vincristine sulfate liposome injection 1.98 mg/m^2 (Experimental): Treatment with the combination of rituximab, bendamustine and vincristine sulfate liposome injection will be repeated every 4 weeks for a maximum of 6 cycles. Dose-limiting toxicities will be evaluated during the first cycle of therapy.
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Vincristine sulfate liposome injection
- Vincristine sulfate liposome injection 2.04 mg/m^2 (Experimental): Treatment with the combination of rituximab, bendamustine and vincristine sulfate liposome injection will be repeated every 4 weeks for a maximum of 6 cycles. Dose-limiting toxicities will be evaluated during the first cycle of therapy.
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Vincristine sulfate liposome injection
- Vincristine sulfate liposome injection 2.10 mg/m^2 (Experimental): Treatment with the combination of rituximab, bendamustine and vincristine sulfate liposome injection will be repeated every 4 weeks for a maximum of 6 cycles. Dose-limiting toxicities will be evaluated during the first cycle of therapy.
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Vincristine sulfate liposome injection
- Vincristine sulfate liposome injection 2.14 mg/m^2 (Experimental): Treatment with the combination of rituximab, bendamustine and vincristine sulfate liposome injection will be repeated every 4 weeks for a maximum of 6 cycles. Dose-limiting toxicities will be evaluated during the first cycle of therapy.
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Vincristine sulfate liposome injection
- Vincristine sulfate liposome injection 2.19 mg/m^2 (Experimental): Treatment with the combination of rituximab, bendamustine and vincristine sulfate liposome injection will be repeated every 4 weeks for a maximum of 6 cycles. Dose-limiting toxicities will be evaluated during the first cycle of therapy.
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Vincristine sulfate liposome injection
- Vincristine sulfate liposome injection 2.22 mg/m^2 (Experimental): Treatment with the combination of rituximab, bendamustine and vincristine sulfate liposome injection will be repeated every 4 weeks for a maximum of 6 cycles. Dose-limiting toxicities will be evaluated during the first cycle of therapy.
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Vincristine sulfate liposome injection
- Vincristine sulfate liposome injection 2.24 mg/m^2 (Experimental): Treatment with the combination of rituximab, bendamustine and vincristine sulfate liposome injection will be repeated every 4 weeks for a maximum of 6 cycles. Dose-limiting toxicities will be evaluated during the first cycle of therapy.
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Vincristine sulfate liposome injection

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 I.V. on Day 1 of each cycle
  Other Names: Rituxan, anti-CD20 antibody
Drug: Bendamustine — 90 mg/m2 I.V. on Day 1 and 2 of each cycle
  Other Names: Treanda
Drug: Vincristine sulfate liposome injection — Dose per dose escalation protocol, I.V. on Day 2 of each cycle
  Other Names: Marqibo

SUMMARY:
This study evaluates addition of Vincristine Sulfate Liposome Injection (Marqibo®) to the standard regimen of Bendamustine and Rituximab in adult patients with indolent B-cell lymphoma. This is a dose-escalation study.

DETAILED DESCRIPTION:
Bendamustine-rituximab is a standard chemotherapy regimen for treatment of many indolent B-cell lymphomas, but most patients experience a recurrence of the lymphoma. Vincristine sulfate has been a traditional component of chemotherapy regimens in non-Hodgkin lymphoma and it is possible that adding it to the bendamustine-rituximab regimen might provide a better quality of remissions or longer duration of remissions with acceptable toxicity.

This is a phase 1, single-center, open-label, single-arm trial in patients with indolent B-cell non-Hodgkin lymphoma otherwise appropriate for bendamustine-rituximab as initial or subsequent line of therapy. Patients will receive the of rituximab and bendamustine in combination with escalating doses of vincristine sulfate liposome injection (Marqibo®). The objective of this study is to assess safety of this combination by establishing the maximum tolerated dose of vincristine sulfate liposome injection (Marqibo®) in the combination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed indolent B-cell non-Hodgkin lymphoma.
* Radiological measurable disease.
* Previous treatment for lymphoma is allowed, with the exception of use of bendamustine within 6 months or any prior use of vincristine sulfate liposome injection
* Eastern Cooperative Oncology Group performance status 0 or 1;
* Life expectancy of at least 6 months;
* Adequate organ and marrow function;
* Women of child-bearing potential and men must agree to use adequate contraception.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of allergic reactions attributed to any drug used in the study.
* Any lymphoma-directed therapy within 4 weeks.
* Any prior treatment with vincristine sulfate liposome injection.
* Prior treatment with bendamustine or vincristine sulfate within 180 days of enrollment.
* Patients who are receiving any other investigational agents with the exception of endocrine therapy for breast or prostate cancer.
* Central nervous system involvement.
* Peripheral sensory or motor neuropathy.
* History of a demyelinating condition.
* Positive test for the Human Anti-Chimeric Antibody (HACA).
* Patients receiving any medications or substances that are strong inhibitors or inducers of Cytochrome P450, family 3, subfamily A (CYP3A) enzyme are ineligible.
* Uncontrolled intercurrent illness.
* Prisoners.
* Pregnant or breast-feeding women.
* Known Human Immunodeficiency Virus (HIV) or active Hepatitis B infection
* Any prior or active cancer, which in the opinion of the investigator would preclude safe participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2020-08-22 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Olszewski, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital and The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ollila T, Butera J, Egan P, Reagan J, Thomas A, Yakirevich I, MacKinnon K, Margolis J, McMahon J, Rosati V, Olszewski AJ. Vincristine Sulfate Liposome Injection with Bendamustine and Rituximab as First-Line Therapy for B-Cell Lymphomas: A Phase I Study. Oncologist. 2022 Jul 5;27(7):532-e542. doi: 10.1093/oncolo/oyab079. PMID 35641232

RESULTS

PARTICIPANT FLOW:
Groups:
- Vincristine Sulfate Liposome Injection: 1.8 mg/m^2; Vincristine Sulfate Liposome Injection: 1.95 mg/m^2; Vincristine Sulfate Liposome Injection: 1.98 mg/m^2; Vincristine Sulfate Liposome Injection: 2.04 mg/m^2; Vincristine Sulfate Liposome Injection: 2.10 mg/m^2; Vincristine Sulfate Liposome Injection: 2.14 mg/m^2; Vincristine Sulfate Liposome Injection: 2.19 mg/m^2; Vincristine Sulfate Liposome Injection: 2.22 mg/m^2; Vincristine Sulfate Liposome Injection: 2.24 mg/m^2: Treatment with the combination of rituximab, bendamustine and vincristine sulfate liposome injection will be repeated every 4 weeks for a maximum of 6 cycles. Dose-limiting toxicities will be evaluated during the first cycle of therapy.
  Rituximab: 375 mg/m2 I.V. on Day 1 of each cycle
  Bendamustine: 90 mg/m2 I.V. on Day 1 and 2 of each cycle
  Vincristine sulfate liposome injection: Dose per dose escalation protocol, I.V. on Day 2 of each cycle
Period: Overall Study
Arm/Group | Vincristine Sulfate Liposome Injection: 1.8 mg/m^2 | Vincristine Sulfate Liposome Injection: 1.95 mg/m^2 | Vincristine Sulfate Liposome Injection: 1.98 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.04 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.10 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.14 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.19 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.22 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.24 mg/m^2
Started | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — 1 subject removed from study before any treatment due to temporary unavailability of study drug | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vincristine Sulfate Liposome Injection: 1.95 mg/m^2; Vincristine Sulfate Liposome Injection: 1.98 mg/m^2; Vincristine Sulfate Liposome Injection: 2.04 mg/m^2; Vincristine Sulfate Liposome Injection: 2.10 mg/m^2; Vincristine Sulfate Liposome Injection: 2.14 mg/m^2; Vincristine Sulfate Liposome Injection: 2.19 mg/m^2; Vincristine Sulfate Liposome Injection: 2.22 mg/m^2; Vincristine Sulfate Liposome Injection: 2.24 mg/m^2: Treatment with the combination of rituximab, bendamustine and vincristine sulfate liposome injection will be repeated every 4 weeks for a maximum of 6 cycles. Dose-limiting toxicities will be evaluated during the first cycle of therapy.
- Total: Total of all reporting groups
Arm/Group | Vincristine Sulfate Liposome Injection: 1.8 mg/m^2 | Vincristine Sulfate Liposome Injection: 1.95 mg/m^2 | Vincristine Sulfate Liposome Injection: 1.98 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.04 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.10 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.14 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.19 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.22 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.24 mg/m^2 | Total
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 7
  >=65 years | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 4
Age, Continuous [Mean (Full Range); unit: years] | 70 [66 to 74] | 40 [40 to 40] | 75 [75 to 75] | 69 [62 to 76] | 58 [58 to 58] | 61 [61 to 61] | 54 [54 to 54] | 57 [57 to 57] | 39 [39 to 39] | 60 [39 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 6
  Male | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 2 | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 2 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 8
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: Determined as the median of the marginal posterior distribution using data from all available patients
Time Frame: Up to 6 cycles of treatment (approximately 6 months)
Measure: Number; unit: mg/m^2
Groups:
- Dose-escalation Cohort: Treatment with the combination of rituximab, bendamustine and vincristine sulfate liposome injection will be repeated every 4 weeks for a maximum of 6 cycles. Dose-limiting toxicities will be evaluated during the first cycle of therapy.
  Rituximab: 375 mg/m2 I.V. on Day 1 of each cycle
  Bendamustine: 90 mg/m2 I.V. on Day 1 and 2 of each cycle
  Vincristine sulfate liposome injection: Dose per dose escalation protocol, I.V. on Day 2 of each cycle
Arm/Group | Dose-escalation Cohort
Number analyzed (Participants) | 10
mg/m^2 | 2.24

2. Secondary Outcome: Number of Participants Who Completed Six Cycles of Study Treatment
Time Frame: Up to 6 cycles of treatment (approximately 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Vincristine Sulfate Liposome Injection: 1.8 mg/m^2 | Vincristine Sulfate Liposome Injection: 1.95 mg/m^2 | Vincristine Sulfate Liposome Injection: 1.98 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.04 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.10 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.14 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.19 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.22 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.24 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1
Participants | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1

3. Secondary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 6 cycles of treatment (approximately 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Vincristine Sulfate Liposome Injection: 1.8 mg/m^2 | Vincristine Sulfate Liposome Injection: 1.95 mg/m^2 | Vincristine Sulfate Liposome Injection: 1.98 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.04 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.10 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.14 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.19 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.22 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.24 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1
Participants
  Complete Response | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
  Partial Response | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
  Stable Disease | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Complete Response Rate
Description: The number of patients achieving complete response during treatment on study
Time Frame: Up to 6 cycles of treatment (approximately 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Vincristine Sulfate Liposome Injection 1.8 mg/m^2 | Vincristine Sulfate Liposome Injection 1.95 mg/m^2 | Vincristine Sulfate Liposome Injection 1.98 mg/m^2 | Vincristine Sulfate Liposome Injection 2.04 mg/m^2 | Vincristine Sulfate Liposome Injection 2.10 mg/m^2 | Vincristine Sulfate Liposome Injection 2.14 mg/m^2 | Vincristine Sulfate Liposome Injection 2.19 mg/m^2 | Vincristine Sulfate Liposome Injection 2.22 mg/m^2 | Vincristine Sulfate Liposome Injection 2.24 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1
Participants | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the date the subject signed the informed consent form for the trail until the end of study visit, approximately 6 months.
Groups:
- Vincristine Sulfate Liposome Injection: 2.1 mg/m^2; Vincristine Sulfate Liposome Injection: 2.14 mg/m^2; Vincristine Sulfate Liposome Injection: 2.19 mg/m^2; Vincristine Sulfate Liposome Injection: 2.22 mg/m^2; Vincristine Sulfate Liposome Injection: 2.24 mg/m^2: Treatment with the combination of rituximab, bendamustine and vincristine sulfate liposome injection will be repeated every 4 weeks for a maximum of 6 cycles. Dose-limiting toxicities will be evaluated during the first cycle of therapy.
  Rituximab: 375 mg/m2 I.V. on Day 1 of each cycle
  Bendamustine: 90 mg/m2 I.V. on Day 1 and 2 of each cycle
  Vincristine sulfate liposome injection: Dose per dose escalation protocol, I.V. on Day 2 of each cycle
Arm/Group | Vincristine Sulfate Liposome Injection: 1.8 mg/m^2 | Vincristine Sulfate Liposome Injection: 1.95 mg/m^2 | Vincristine Sulfate Liposome Injection: 1.98 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.04 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.1 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.14 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.19 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.22 mg/m^2 | Vincristine Sulfate Liposome Injection: 2.24 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/2 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 1/2 | 0/1 | 1/1 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 2/2 | 1/1 | 1/1 | 1/1 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vincristine Sulfate Liposome Injection: 1.8 mg/m^2 (N=1) | Vincristine Sulfate Liposome Injection: 1.95 mg/m^2 (N=1) | Vincristine Sulfate Liposome Injection: 1.98 mg/m^2 (N=1) | Vincristine Sulfate Liposome Injection: 2.04 mg/m^2 (N=2) | Vincristine Sulfate Liposome Injection: 2.1 mg/m^2 (N=1) | Vincristine Sulfate Liposome Injection: 2.14 mg/m^2 (N=1) | Vincristine Sulfate Liposome Injection: 2.19 mg/m^2 (N=1) | Vincristine Sulfate Liposome Injection: 2.22 mg/m^2 (N=1) | Vincristine Sulfate Liposome Injection: 2.24 mg/m^2 (N=1)
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thromboembolic Event (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vincristine Sulfate Liposome Injection: 1.8 mg/m^2 (N=1) | Vincristine Sulfate Liposome Injection: 1.95 mg/m^2 (N=1) | Vincristine Sulfate Liposome Injection: 1.98 mg/m^2 (N=1) | Vincristine Sulfate Liposome Injection: 2.04 mg/m^2 (N=2) | Vincristine Sulfate Liposome Injection: 2.1 mg/m^2 (N=1) | Vincristine Sulfate Liposome Injection: 2.14 mg/m^2 (N=1) | Vincristine Sulfate Liposome Injection: 2.19 mg/m^2 (N=1) | Vincristine Sulfate Liposome Injection: 2.22 mg/m^2 (N=1) | Vincristine Sulfate Liposome Injection: 2.24 mg/m^2 (N=1)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chills (General disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fever (General disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 1 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1
Neck edema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Weight loss (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
White blood cell decreased (Investigations) | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT02257242/Prot_SAP_ICF_000.pdf